CLINICAL TRIAL: NCT07167901
Title: The Impact of Free Gingival Grafts on Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Principal Investigator, Serap Karakış Akcan, Asst. Prof, Istanbul Gelisim University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-16-79
Record Dates: First submitted 2025-07-09; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Free Gingival Graft; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: parallel clinical prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prosthetically restored teeth (Experimental): Prosthetically restored teeth will also be included in this group. Free gingival graft surgery will be performed
  Interventions: Procedure: Free Gingival Graft
- Non-restored teeth (Experimental): Non-restored teeth will also be included in this group. Free gingival graft surgery will be performed
  Interventions: Procedure: Free Gingival Graft

INTERVENTIONS:
Procedure: Free Gingival Graft — All patients will undergo free gingival graft surgery by the same surgeon using the same surgical protocol.

SUMMARY:
This study compares the effects of free gingival graft (FGG) surgery on prosthetically restored and non-restored teeth regarding patients' oral quality of life using various scales. Patients with insufficient attached gingiva who are indicated for free gingival graft surgery will be included in this study. We will collect demographic data, including age, gender for all patients who meet the inclusion criteria. Prior to the surgery, all patients will have their oral periodontal indices and their scores on the Oral Health Impact Profile-14 (OHIP-14) recorded. All patients will undergo free gingival graft surgery using the same surgical technique, and we will record operation details such as graft dimensions and the location of the recipient bed. The OHIP-14 will be completed three times: once one day, one week, and again one month after the surgery. Additionally, a satisfaction questionnaire will be administered one month post-operation, and a visual analog scale (VAS) for pain will be collected during one week after the surgery. Following statistical analysis of the collected data, we will report on the impact of the free gingival graft surgery on oral health-related quality of life. The distribution of OHIP-14 scores, satisfaction survey results, and VAS pain scale data will be analyzed in relation to demographic characteristics and their association with surgical data.

DETAILED DESCRIPTION:
This clinical study is designed to evaluate the impact of free gingival graft (FGG) surgery on oral health-related quality of life in patients with insufficient attached gingiva. Participants will be recruited from the Departments of Periodontology at Istanbul Gelişim University and Kütahya Health Sciences University.

All participants will receive phase I periodontal treatment and oral hygiene instructions prior to surgery. After a four-week healing period, FGG surgery will be performed using a standardized surgical technique. Surgical data, including graft dimensions and recipient site location, will be recorded during the procedure.

Participants will be categorized into two groups based on the presence or absence of prosthetic restoration on the treated tooth:

Group 1: Non-restored teeth

Group 2: Prosthetically restored teeth

Clinical periodontal indices will be assessed at baseline and postoperatively. Oral health-related quality of life will be evaluated using the OHIP-14 questionnaire administered at baseline, one day, one week, and one month following surgery. Patient-reported outcomes will include a satisfaction questionnaire at one month and a visual analog scale (VAS) for postoperative pain during the first week. The number of analgesics consumed will also be recorded.

The primary objective is to compare changes in OHIP-14 scores between groups over time. Secondary outcomes include postoperative pain, patient satisfaction, and the association of clinical and surgical parameters with quality of life measures.

Data will be analyzed using descriptive and inferential statistics. Normality of distribution will be tested, and comparisons between repeated measures and groups will be conducted with appropriate parametric or non-parametric tests. Correlation analyses will be performed to examine relationships between clinical, surgical, and patient-reported variables. The calculated sample size is 49 participants, accounting for potential dropouts.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* The patient does not have any systemic disease
* The patient is cooperative
* Patients with keratinized mucosa deficiency or insufficiency (less than 1 mm)

Exclusion Criteria:

* regnant and breastfeeding patients
* Mentally retarded patients
* Patients who smoke more than 10 cigarettes per day
* Patients with bleeding disorders or anticoagulant medication use
* Patients who use medications that suppress the immune system or impair healing
* Patients who do not answer the questions in a timely manner and cannot cooperate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Oral health impact profile- 14 Scale | Before FGG surgery and After 1 day, 1 week, and 1 month
  Oral health impact profile- 14 Scale OHIP-14 questionnaire: OHIP-14 consists of 14 questions and Likert scale is used (0=Never, 1=Rarely, 2=Sometimes, 3=Frequently and 4=Always). In the evaluation of OHIP-14, scoring is done separately in 7 categories under the main titles of functional limitation, physical pain, psychological discomfort, physical disability, psychological disability and handicap and the total score obtained by the sum of all these category scores
Satisfaction questionnaire | 1 month after the sugery
  The satisfaction survey consists of 13 questions and is answered as yes or no. The patient's level of satisfaction with the treatment will be assessed with a 13-question survey asked 1 month after the Free Gingival Graft treatment.

SECONDARY OUTCOMES:
VAS pain scale | 1 week during after the surgery
  VAS VISUAL ANALOG SCALE (VAS) PAIN SCALE: The post-operative pain levels of the patients will be evaluated with the VAS pain scale. The pain felt will be marked on the VAS pain scale. On the horizontal scale, 0 means no pain, and 100 means unbearable pain.
Number of painkillers used | 1 week during after the surgery
  Number of painkillers used
Clinical periodontal index | Before FGG surgery and 1 month after the sugery
  Clinical periodontal measurements are given below. Plaque index Gingival index Bleeding index on probing Pocket depth Clinical attachment level Keratinized gingival width
Operational data | On the surgery
  Graft width (mm) Graft length (mm) Graft thickness(mm) Graft volume (Graft width x Graft length x Graft thickness ) Recipient bed location (maxilla-mandible, anterior-posterior)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Gelisim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It can be shared if the responsible researcher is contacted.